CLINICAL TRIAL: NCT03836469
Title: Retrospective Epidemiological Study of Locally Advanced Non Small Cell Lung Cancer Patients in Brazil
Acronym: RELANCE
Status: Completed | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: LACOG 0118
Record Dates: First submitted 2019-02-08; First posted 2019-02-11 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Lung Cancer, Non-small Cell
Keywords: Lung cancer; Non-small cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
RELANCE is a large multi-institutional study that aims to retrospectively collect information about diagnostic, treatment and outcome of patients diagnosed with locally advanced NSCLC in Brazil. It is hypothesized that there is a great heterogeneity in treatment patterns owing to inequities in access to adequate staging methods, optimal treatment and multidisciplinary teams in Brazil.

DETAILED DESCRIPTION:
RELANCE study will collect sociodemographic and clinical data of patients diagnosed with locally advanced NSCLC in the period of January 2015 and Jun 2019 in the participating institutions. Socio-demographic characteristics, clinicopathological features, treatments patterns and outcomes will be recovered from medical charts. Disease status and survival data will be collected up to the last date of follow-up June 2021.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older;
2. Histologically or cytological diagnosis of NSCLC in the period of January 2015 to December 2016;
3. Locally Advanced NSCLC defined as clinical stage IIIA and IIIB according to 7th Edition TNM Staging System;
4. Any NSCLC histological subtype and molecular mutation;
5. Any Eastern Cooperative Oncology Group (ECOG) Performance Status (0 to 4) at diagnosis;
6. Patients assigned by treating physician to any therapy or palliative care;
7. Access to patient medical chart for data collection.

Exclusion Criteria:

1. Small cell lung cancer and non-invasive NSCLC;
2. Synchronic NSCLC or second primary tumour in the last 5 years (except non-melanoma skin cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with stage IIIA or IIIB NSCLC in the period of January 2015 to December 2016.
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to June 30, 2018
  defined as time from diagnosis to death of any cause;

SECONDARY OUTCOMES:
Progression free survival | Up to June 30, 2018
  defined as time from any line of treatment to progression of the disease or death of any cause
Time to next treatment | Up to June 30, 2018
  defined as time from start of the any treatment to the beginning of a second therapy

CONTACTS AND LOCATIONS:
Overall Officials: Vladmir Cláudio Cordeiro de Lima, Principal Investigator — Latin American Cooperative Oncology Group
Locations (1):
- AC Camargo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No